CLINICAL TRIAL: NCT00017017
Title: A Phase I/II Trial fo Intravenous CT-2103 in Patients With Recurrent Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Carcinoma
Brief Title: CT-2103 in Treating Patients With Recurrent Ovarian Epithelial or Fallopian Tube Cancer or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CTI-1071; MSKCC-01024; CDR0000068642 (Registry Identifier: PDQ (Physician Data Query)); NCI-G01-1947
Record Dates: First submitted 2001-06-06; First posted 2003-11-13 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2009-12

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — paclitaxel poliglumex

INTERVENTIONS:
Drug: paclitaxel poliglumex

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I/II trial to study the effectiveness of CT-2103 in treating patients who have recurrent ovarian epithelial or fallopian tube cancer or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate and time to treatment failure in patients with recurrent ovarian epithelial, fallopian tube, or primary peritoneal carcinoma treated with CT-2103.
* Determine the tolerability and safety of the previously established dose and schedule of CT-2103 in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive CT-2103 IV over 10 minutes on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

If no more than 1 of the first 6 patients experience dose-limiting toxicity, then the remaining patients receive a higher dose of CT-2103.

Patients are followed between 1-3 months and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, fallopian tube, or primary peritoneal carcinoma

  * Recurrent disease following prior initial therapy with platinum-based regimen

    * No more than 2 prior cytotoxic chemotherapy regimens for recurrent disease
    * No more than 1 prior non-platinum, non-taxane regimen
* At least 1 site of radiographically measurable disease AND/OR
* CA-125 levels at least 50% above upper limits of normal for a minimum of 2 samples

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT less than 1.5 times ULN
* Alkaline phosphatase less than 1.5 times ULN

Renal

* Creatinine no greater than 1.5 mg/dL

Other

* No unresolved, pre-existing grade 2 or greater neurotoxicity from prior treatment with neurotoxic drugs
* No active uncontrolled infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 weeks after study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 4 weeks since prior immunotherapy and recovered

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy and recovered

Endocrine therapy

* At least 4 weeks since prior endocrine therapy and recovered

Radiotherapy

* At least 4 weeks since prior radiotherapy (except for palliative reasons) and recovered

Surgery

* Not specified

Other

* At least 4 weeks since other prior investigational drugs and recovered

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-02; Primary Completion 2003-02 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sabbatini, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States